CLINICAL TRIAL: NCT07347158
Title: Effectiveness of Health Education as a Nursing Intervention in Improving Quality of Life and Reducing Symptoms of Anxiety and Depression in Ostomy Patients Following Digestive Surgery: A Quasi-Experimental Study.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Collaborators: Hospital Clínico Universitario de Santiago de Compostela (Unknown)
Responsible Party: Principal Investigator, Tomás Mendoza Caamaño, Tomás Mendoza Caamaño, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024-389
Record Dates: First submitted 2025-12-04; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Colon Cancer; Inflamatory Bowel Disease (Crohn's and Ulcerative Colitis); Colitis Ulcerative
Keywords: ostomy; quality of life; anxiety; depression; Nursing care; Health education; stoma care
MeSH Terms: conditions — Colonic Neoplasms; Colitis, Ulcerative; Anxiety Disorders; Depression; Health Education

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health education by virtual and smart-glasses (Experimental): Health education (emotional care, mindfulness, jacobson, quality of life, social, sexual, ...). Method: psicosocial/holistic
  Interventions: Other: Health Education
- Control (No Intervention)

INTERVENTIONS:
Other: Health Education — Session 1 (60 minutes) Patient Knowledge Assessment: Review understanding of ostomy care, including nutrition, device management, and early identification of stoma/skin complications.
  Feedback and Support: Address gaps in knowledge based on ostomy consultations. Skills Workshop: Build confidence and self-efficacy in daily care, reducing anxiety about complications.
  Session 2 (60 minutes) Mental Health and Quality of Life: Explain the link between ostomy and mental health; identify and manage anxiety/depression symptoms; promote healthy habits and social integration.
  Mindfulness and Stress Management: Teach breathing and relaxation techniques to manage stress and improve body acceptance.
  Guided Visualization: Focus on acceptance and confidence building. Action Plan: Summarize techniques and encourage regular practice. Session 3 Healthy Habits: Nutrition, exercise, rest, and stress management. Social Integration: Communication, participation, and support networks. Closing: Summary, resou
  Arms: Health education by virtual and smart-glasses

SUMMARY:
The proposed project is a prospective quasi-experimental study to be conducted at the Ostomy Clinic of the University Hospital Complex of Santiago de Compostela. The primary objective is to evaluate the effectiveness of health education as a nursing intervention in reducing anxiety and depression and improving the quality of life of ostomy patients following digestive surgery. The study will focus on adult patients who have undergone an elimination ostomy, excluding terminal patients and those with cognitive impairments.

The study involves clinical follow-up of patients from hospital admission to several months after completing the health education program. Validated scales will be used to measure quality of life, anxiety, and depression. The intervention will consist of health education workshops and continuous follow-up by specialized nursing staff.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Patients with digestive ostomies, either permanent or temporary ostomies lasting more than 6 months, attending ostomy consultations.
* Volunteers with permanent digestive ostomies from the Santiago and Barbanza healthcare area.
* Patients who agree to participate in the study.

Exclusion Criteria:

* Terminal patients
* Patients with cognitive impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-03-04 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory | Baseline and at 3 months
  Beck Depression Inventory
36-Item Short Form Health Survey | Baseline and at 3 months
  36-Item Short Form Health Survey
Beck anxiety inventory | Baseline and at 3 months
  Beck anxiety inventory

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-26): https://cdn.clinicaltrials.gov/large-docs/58/NCT07347158/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-26): https://cdn.clinicaltrials.gov/large-docs/58/NCT07347158/ICF_001.pdf